CLINICAL TRIAL: NCT07152431
Title: FATE-CD: A Prospective Cohort Observational Study Investigating the Role of Fibrosis Activity in Crohn's Disease
Brief Title: Fibrosis Associated Protein Inhibitor (FAPI) Radiotracer-based Imaging to Identify Fibrotic Intestinal Crohn's Disease
Acronym: FATE-CD
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 332586
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
Keywords: fibrosis
MeSH Terms: conditions — Crohn Disease; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's Disease (CD) is a chronic inflammatory condition that can affect any part of the intestine and currently has no cure. It affects 6.8 million people worldwide with UK healthcare costs in excess of £1 billion per year. Recent data suggests that the despite significant progress in treatments over the last 2 decades to help control disease, up to half of patients still develop progressive bowel scarring that require surgery and up to 70% needing surgery within 10-20 years from diagnosis. Unfortunately this is not a cure and some still require repeat surgery. These features have a devastating impact on an individual including education, work and social life. All our current treatments focus on resolving inflammation but there are no treatments targeting fibrosis, its activity and its progression. A major hurdle in our progress towards anti-fibrotic treatments and advancing care in CD has been our inability to identify bowel scarring accurately using non-invasive tests; this being critical in developing new treatments that prevent permanent bowel damage.

We are also unable to identify early stage scarring (fibrosis) and once established we are unable to differentiate between different stages of scarring severity.

The investigators aim to investigate a novel method that can identify early scarring and track progressive bowel damage by tracking cells that cause fibrosis. In this study the investigators will use a 'dye', also known as fibrosis associated protein inhibitor (FAPI), that tracks scarring and its activity in the intestine. The presence and amount of FAPI within an area of scarring can be detected using our current imaging tests (positron emission tomography and Computer Tomography imaging: PET/CT). If successful, this study will be the first method for detecting scarring activity in CD and have the potential to revolutionise care for this condition and facilitate new drug development to halt the processing of scarring (fibrosis) and improve the outcomes for patients with CD.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease with ileal involvement (including those with disease recurrence in the neo-terminal ileum) due to commence biologics.

Exclusion Criteria:

* Inability or unwilling to give informed consent.

  * History of claustrophobia or feeling of inability to tolerate supine position for the PET/MRI or PET/CT scans.
  * Impaired renal function with eGFR of <30 mL/min/1.73m2
  * Women who are pregnant or breastfeeding. Pregnancy test will be performed in all women of childbearing age
  * Contrast allergy
  * Contraindication to MRI (e.g. metallic implant or severe claustrophobia)
  * Significant mental health conditions that will impair the ability to consent or affect their ability to take part in the study
  * Patients with colonic disease only with no ileal or small bowel involvement.
  * Contraindications (Glaucoma and/or ischaemic heart disease) or allergy (eg:

anaphylaxis) to buscopan use.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Crohn's disease and small bowel involvement
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Fibrosis activity | 36 months
  To establish and quantify the intestinal fibrosis activity in patients with active fibrostenosing Crohn's disease phenotype (Montreal B2) and assess its utility in predicting fibrosis progression over time

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No